CLINICAL TRIAL: NCT00004759
Title: Phase III Randomized, Double-Blind Study of Methylprednisolone by 24- Versus 48-Hour Infusion Versus Tirilazad for Acute Spinal Cord Injury
Brief Title: Methylprednisolone Given by 24-Hour or 48-Hour Infusion Versus Tirilazad for Acute Spinal Cord Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: Yale University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11692; YALESM-5908
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2008-09-10 (Estimated); Status verified 2008-09

CONDITIONS: Spinal Cord Injury
Keywords: environmental/toxic disorders; neurologic and psychiatric disorders; rare disease; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Methylprednisolone; tirilazad

INTERVENTIONS:
Drug: methylprednisolone
Drug: tirilazad

SUMMARY:
OBJECTIVES:

I. Compare the efficacy and safety of 24- versus 48-hour infusion of methylprednisolone (MePRDL) versus tirilazad for patients with acute spinal cord injury.

II. Compare neurologic recovery following 24- and 48-hour MePRDL infusions.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a randomized, double-blind study. Patients are stratified by participating institution.

Patients are randomly assigned to 1 of 3 treatment groups within 6 hours of injury. Treatment begins within 2 hours of randomization.

One group receives a 24-hour methylprednisolone (MePRDL) infusion: a loading dose followed in 45 minutes by a 23-hour continuous infusion. A placebo for tirilazad is also administered.

A second group receives the same MePRDL loading dose but the continuous infusion is maintained for 48 hours. A placebo for tirilazad is also administered.

A third group receives a 48-hour infusion of tirilazad with an initial bolus dose of MePRDL. Eight additional doses of tirilazad are administered by intravenous push. The MePRDL loading dose may be omitted for patients who received a prestudy MePRDL dose.

Patients are followed at 72 hours, 6 weeks, 6 months, and 1 year after the injury.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Acute spinal cord injury; diagnosis confirmed by study physician using National Acute Spinal Cord Injury Study neurologic exam

Glasgow Coma Score greater than 9

Randomization within 6 hours of injury required; treatment must begin within 8 hours of injury

No root involvement only; no cauda equina only

--Prior/Concurrent Therapy--

Methylprednisolone bolus (20-40 mg/kg) prior to hospital admission allowed

--Patient Characteristics--

Hematopoietic: No hematologic contraindication to protocol therapy

Cardiovascular: No vascular contraindication to protocol therapy

Other: No diabetes; No gunshot wound; No gastrointestinal bleeding; No life-threatening co-morbidity; No other medical contraindication to protocol therapy; No pregnant women; No patients under indictment or incarcerated; No conditions that would complicate follow-up, e.g.: out-of-state residency or illegal alien status

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 497
Dates: Start 1991-12; Primary Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bracken, Study Chair — Yale University

REFERENCES:
- [Background] Bracken MB, Shepard MJ, Holford TR, Leo-Summers L, Aldrich EF, Fazl M, Fehlings MG, Herr DL, Hitchon PW, Marshall LF, Nockels RP, Pascale V, Perot PL Jr, Piepmeier J, Sonntag VK, Wagner F, Wilberger JE, Winn HR, Young W. Methylprednisolone or tirilazad mesylate administration after acute spinal cord injury: 1-year follow up. Results of the third National Acute Spinal Cord Injury randomized controlled trial. J Neurosurg. 1998 Nov;89(5):699-706. doi: 10.3171/jns.1998.89.5.0699. PMID 9817404
- [Background] Bracken MB, Shepard MJ, Holford TR, Leo-Summers L, Aldrich EF, Fazl M, Fehlings M, Herr DL, Hitchon PW, Marshall LF, Nockels RP, Pascale V, Perot PL Jr, Piepmeier J, Sonntag VK, Wagner F, Wilberger JE, Winn HR, Young W. Administration of methylprednisolone for 24 or 48 hours or tirilazad mesylate for 48 hours in the treatment of acute spinal cord injury. Results of the Third National Acute Spinal Cord Injury Randomized Controlled Trial. National Acute Spinal Cord Injury Study. JAMA. 1997 May 28;277(20):1597-604. PMID 9168289